CLINICAL TRIAL: NCT05434429
Title: Evaluating the Effectiveness of a Smartphone App to Reduce Craving and Lapse Risk in Problematic Behaviors and Substance Use
Brief Title: Mobile Health for Problematic Behaviors and Substance Use
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: PredictWatch (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/002A
Record Dates: First submitted 2022-06-22; First posted 2022-06-28 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Addiction; Behavioral Addiction; Nicotine Addiction; Nicotine Dependence; Cannabis Dependence
Keywords: Addiction; mHealth; mobile app; Cannabis; Nicotine; Behavioral Addiction
MeSH Terms: conditions — Behavior, Addictive; Tobacco Use Disorder; Marijuana Abuse

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants have access to short-term and long-term interventions.
  Interventions: Other: mobile application
- Control (No Intervention): Given access to all interventions at the end of the 5 weeks of the trial.

INTERVENTIONS:
Other: mobile application — Participants in the intervention group are able to access the intervention materials 5 days after enrollment. Two main self-guided intervention modules are available. Short-term self-guided intervention module include mainly audio-guided sessions on gratitude, thoughts management, auto-empathy, and relaxation. Moreover, there based on breath relaxation exercises, craving management, and motivation to change. Long-term self-guided intervention module include CBT-based interventions, meditations, mindfulness, and journaling.
  Arms: Intervention

SUMMARY:
The aim of the study is to evaluate the effectiveness of long-term and short-term app-based self-guided psychological interventions to reduce craving and lapse risk in problematic behaviors (compulsive sex, pornography, overeating, gaming, gambling) and substance use (cannabis, nicotine). Participants are randomly assigned to either the intervention group or the control. Participants in the intervention group have access to short-term and long-term interventions, whereas those in the control group only have access to the weekly ecological momentary assessment reports. Participants in the intervention group are able to access the intervention materials 5 days after enrollment and receive weekly ecological momentary assessment reports. Those in the control group will be granted access to all intervention materials after five weeks following study enrollment. A questionnaire battery assessments is administered (1) at baseline in the first week following onboarding in; (2) after 5 weeks; (3) after six months. In addition, longitudinal data on several variables related to craving and lapse risk are collected daily using ecological momentary assessment

DETAILED DESCRIPTION:
The aim of the study is to evaluate the effectiveness of long-term and short-term app-based self-guided psychological interventions to reduce craving and lapse risk in problematic behaviors and substance use.

Two main self-guided intervention modules are available. Short-term self-guided intervention module include mainly audio-guided sessions on gratitude, thoughts management, auto-empathy, and relaxation. Moreover, there based on breath relaxation exercises, craving management, and motivation to change Long-term self-guided intervention module include CBT-based interventions, meditations, mindfulness, and journaling.

Participants are recruited via newsletters, local and nation-wide advertisements, as well as through social media. The study is conducted via a mobile application "Nałogometr", freely available to participants. We recruit people from the general population residing in Poland.

To compare the effectiveness of mobile app-based self-guided psychological interventions, study participants are randomly assigned to either the intervention group or the control.

Experimental conditions are balanced based on multiple variables provided during onboarding: (1) main addiction type; (2) participation in addiction-related therapy; (3) gender; (4) age; (5) addiction severity; (6) abstinence duration.

Participants in the intervention group have access to short-term and long-term interventions, whereas those in the control group only have access to the weekly ecological momentary assessment reports. Participants in the intervention group will be able to access the intervention materials 5 days after enrollment and will receive weekly ecological momentary assessment reports. Those in the control group will be granted access to all intervention materials after five weeks following study enrollment.

Questionnaire battery assessments will take place: (1) at baseline in the first week following onboarding in; (2) after 5 weeks; (3) after six months. In addition, longitudinal data on several variables related to craving and lapse risk will be collected daily using ecological momentary assessment.

ELIGIBILITY:
Inclusion Criteria:

* are at least 18 years of age
* speak Polish fluently
* use either an Android or iOS smartphone

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-06-21 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Lapses rate according to EMA self-report | 5 weeks
  Collected daily via the participant's smartphone; an item asking whether or not the lapse occurred since the last survey (yes / no). The score will be tracked for changes over time.
Craving level according to EMA self-report | 5 weeks
  Collected daily via the participant's smartphone; an item asking how strong is one's urge to use [substance] at the moment on a scale of 0 to 6 (none - incalculable ). The score will be tracked for changes over time.

SECONDARY OUTCOMES:
Binge Eating Disorder Screener-7 | 1 week, 5 weeks, 6 months
  The BEDS-7 screener consists of 7 questions to detect the possibility of the patient having Binge Eating Disorder (BED) (Herman et al., 2016). First, a filter question is asked if the participant experienced at least one episode of excessive overeating during the last 3 months; if answered yes, the next question if about feeling distress from episodes of excessive eating (with possible answers: 'Yes', 'No'), followed by five questions using a Likert-like rating scale ('Never or Rarely', 'Sometimes', 'Often', 'Always'). An answer of 'Yes' to both first two questions with a response of 'Often', 'Always', or 'Sometimes' to questions 3 - 6, and an answer of 'Never or Rarely' or 'Sometimes' to question 7 will yield a result of showing symptoms of BED.
Brief Pornography Screen-PL | 1 week, 5 weeks, 6 months
  Pornography use will be measure with Brief Pornography Screener (BPS) (Kraus et al., 2019), a 5-item, one-dimensional scale. All questions regards to pornography use in last six month and are scored on 0 ('never') to 2 ('very often'). Minimum score is 0 and maximum is 10. Total score 4 and over indicates problematic pornography use.
The Cannabis Use Disorder Identification Test - Revised | 1 week, 5 weeks, 6 months
  Cannabis Use Disorder will be accessed with The Cannabis Use Disorders Identification Test-Revised (CUDIT-R) (Adamson et al., 2010), an eight items one-dimensional scale. Questions from 1 to 7 are scored on a 0 ('never) to 4 ('daily or almost daily') scale, and a question 8 is scored as 0 ('never'), 2 ('Yes, but not in the past 6 months') or 4 ('Yes, during the past 6 months'). A score between 8 and 11 indicates hazardous cannabis use, and scores above 12 points indicate possible cannabis use disorder.
The Fagerstrom Test for Nicotine Dependence | 1 week, 5 weeks, 6 months
  Nicotine dependence was assessed by The Fagerstrom Test for Nicotine Dependence (FTND) (Heatherton et al., 1991). The questionnaire is composed of 6 questions, with varying choices in each question. Each option is accompanied by a number indicating its score for the questionnaire scoring system. The total score is categorized as follows: 0-2 indicates a very low dependence, 3-4 indicates a low dependence, 5-7 indicates a moderate-to-high dependence, lastly, 8+ indicates a very high dependence. In addition, a filter question inquiring if the participant is a user of nicotine products was asked before the questionnaire.
Drug Use Disorders Identification Test | 1 week, 5 weeks, 6 months
  The Drug Use Disorders Identification Test (DUDIT) (Berman et al., 2005) will be used to measure self-report problematic drug use. The DUDIT is an 11-item screening instrument, the first nine items are scored on a 5-point scale (0 - 4 ), and the last two are scored on a 3-point scale (0, 2, and 4, respectively). The overall score is a sum of scores on all items, with a maximum of 44.
  A cut-off of >24 has been used for indexing dependence for both sexes (Berman et al., 2005).
Severity of Dependence Scale | 1 week, 5 weeks, 6 months
  The Severity of Dependence Scale (SDS) (Gossop, et al., 1995) will be used to provide a self-reported measure of psychological aspects of stimulants and alcohol dependence. A five-items, one-dimensional tool has uniform scale for questions 1 - 4 from 0 ('never or almost never') to 3 ('always'). Question 5 has the same scale with different signature where 0 means 'not difficult at all' and 3 means 'impossible'. Score ranging from 0 to 15, where cut-off score depends on user's drug type, while higher values reflect higher dependence.
Compulsive Sexual Behavior Disorder | 1 week, 5 weeks, 6 months
  Compulsive Sexual Behavior Disorder will be accessed with a short version of the Compulsive Sexual Behavior Disorder Scale (CSBDS-19) (Bőthe et al., 2020), including 19 items with possible answers from 1 - strongly disagree to 4 - strongly agree. Tool has five scales: control (items 1,6,11), salience (items 2, 7, 12, relapse (items 3, 8, 13), dissatisfaction (4, 9, 14), and negative consequences (items 5,10,15, 16, 17, 18, 19). The minimum score is 19, and the maximum is 76, with a cut-off of 50 points indicating possible compulsive sexual behavior disorder.
Satisfaction with Life Scale | 1 week, 5 weeks, 6 months
  Participants' satisfaction with their life will be assessed with The Satisfaction With Life Scale (SWLS) (Diener et al., 1985), Polish version from Jankowski (2015). SWLS is a short self-report instrument on which participants indicate their agreement to five statements about life satisfaction on a seven-point Likert scale. A maximum score of 35 can be reached, indicating a high level of life satisfaction.
The Hospital Anxiety Depression Scale | 1 week, 5 weeks, 6 months
  Depression and anxiety will be assessed with Hospital Anxiety and Depression Scale (HADS) (Zigmond and Snaith, 1983; Karakuła et al., 2017), a 14 items two-dimensional tool. Each subscale consists of 7 items, scoring from 0 to 3. For each subscale, scores between 8 and 10 indicate mild depression/anxiety, and scores between 11 and 21 indicate depression/anxiety disorder.
The South Oaks Gambling Screen | 1 week, 5 weeks, 6 months
  Gambling disorder will be masured with South Oaks Gambling Screen (SOGS) (Lessieur, et al., 1987) with 16 items of the one-dimensional tool. The participant is asked to indicate the type of gambling he/she practices at least once in his/her life. The first three questions are qualitative: participants indicated how much money they put at risk at maximum in their life, who from their surroundings tend to gamble, and how they come back the next day to get back. The rest of the items are answered yes/no, and each 'yes' answer is rated as 1 point. The score is calculated as a sum (without questions 1,2,3,12, and 16) with 0 meaning no problem with gambling, 1-4 indicating minor issues with gambling, and scores higher than 4 indicating the risk of pathological gambling.
Internet Gaming Disorder Scale-Short-Form | 1 week, 5 weeks, 6 months
  Gaming disorder was assessed using Internet Gaming Disorder Scale-Short-Form (IGDS9-SF), a 9- items one dimensional tool reflecting nine criteria for Internet Gaming Disorder in DSM-5 (Pontes et al., 2015), Polish version from Schivinski i in. (2018). Items are rated on 5-point scale (1='never', 2= 'rarely', 3='sometimes', 4 = 'often', 5= 'very often') and results can range from a minimum of 9 to a maximum of 45 points, with higher scores indicating higher degree of IGD and a cut-off of 32 (Qin et al., 2020).

CONTACTS AND LOCATIONS:
Locations (1):
- PredictWatch, Bialystok, Poland